CLINICAL TRIAL: NCT03095508
Title: Prospective, Multicenter, Open, Randomized, Parallel, Clinical Study for Comparative Assessment of Efficacy and Safety of Angal S, Topical Spray [Menthol], 0,5 mg + 2 mg / 1 ml (Sandoz d.d., Slovenia), and ANTI-ANGIN® FORMULA, Topical Metered Spray, 0,12 mg + 0,24 mg / Dose (OOO "Valeant", Russia) in Treatment of Patients With Uncomplicated Acute Infectious and Inflammatory Diseases of the Pharynx, Accompanied by a Sore Throat
Brief Title: Clinical Study for Comparative Assessment of Efficacy and Safety of Angal S, Topical Spray and ANTI-ANGIN® FORMULA, Topical Metered Spray in Treatment of Patients With Uncomplicated Acute Infectious and Inflammatory Diseases of the Pharynx, Accompanied by a Sore Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TE_003_ANG_LSP
Record Dates: First submitted 2017-03-24; First posted 2017-03-29 (Actual); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: Sore Throat
Keywords: Angal S; ANTI-ANGIN FORMULA; Sore Throat; no less therapeutic efficacy
MeSH Terms: conditions — Pharyngitis | interventions — Menthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angal S (Arm A) (Experimental): Patients received Angal S, topical spray [Menthol], 0,5 mg + 2 mg (Sandoz d.d., Slovenia), administered as three to five consecutive presses on the actuator button, 6-10 times per day, for a maximum 4 days or until full illness resolution
  Interventions: Drug: Angal S, topical spray [Menthol]
- ANTI-ANGIN® FORMULA (Arm B) (Active Comparator): Patients received ANTI-ANGIN® FORMULA, topical metered spray, 0,12 mg + 0,24 mg (LLC "Valeant", Russia) administered as three to five consecutive presses on the actuator button, 6-10 times per day, for a maximum 4 days or until full illness resolution
  Interventions: Drug: ANTI-ANGIN® FORMULA, topical metered spray

INTERVENTIONS:
Drug: Angal S, topical spray [Menthol] — 0,5 mg + 2 mg (Sandoz d.d., Slovenia), administered as three to five consecutive presses on the actuator button, 6-10 times per day, for a maximum 4 days or until full illness resolution
  Arms: Angal S (Arm A)
Drug: ANTI-ANGIN® FORMULA, topical metered spray — 0,12 mg + 0,24 mg (LLC "Valeant", Russia) administered as one to two consecutive presses on the actuator button, up to 6 times per day, , for a maximum 5 days or until full illness resolution
  Arms: ANTI-ANGIN® FORMULA (Arm B)

SUMMARY:
The purpose of this study was to evaluate no less therapeutic efficacy and safety of the Angal S, topical spray [Menthol], 0,5 mg + 2 mg (Sandoz dd, Slovenia) compared to ANTI-ANGIN® FORMULA, topical metered spray, 0,12 mg + 0,24 mg (LLC "Valeant", Russia) in treatment of patients with uncomplicated acute infectious and inflammatory diseases of the pharynx, accompanied by a sore throat.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent for participation in this clinical study;
* 18 to 45 years old inclusive, male and female;
* Diagnosed uncomplicated acute infectious and inflammatory diseases of the pharynx, accompanied by a sore throat;
* Onset of first symptoms of the uncomplicated acute infectious and inflammatory diseases of the pharynx (pharyngitis and/or tonsillitis) less than 48 hours prior to inclusion into the study; Baseline TSS score (Tonsillopharyngitis Severity Score) ≥ 5 (total score);
* Body temperature 37,5 C (axillary).

Exclusion Criteria:

* Use of analgesics within <12 hours prior to the study start or/and inability to cancel them during the study;
* Use of antibiotics within <48 hours prior to the study start or/and inability to cancel them during the study;
* Use of local therapy (sprays, rinses, lozenges) to pharynx within <12 hours before study start or/and inability to cancel them, besides study medications;
* Use systemic or inhaled corticosteroids within ≤1 months prior to the study start and planned therapy of them during the study (besides skin means);
* Presence of symptoms of primary bacterial pharyngitis or secondary bacterial infection (including fever over 37,5 ° C, the presence of purulent raids in the throat, severe intoxication, leukocytosis, neutrophilia, shift leukocyte left (increasing the percentage of neutrophils sticks appearance younger forms of neutrophils), increased ESR 30 mm/hr).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (4):
- Russia (4):
  - Sandoz Investigational Site, Arkhangelsk
  - Sandoz Investigational Site, Moscow
  - Sandoz Investigational Site, Saint Petersburg
  - Sandoz Investigational Site, Stavropol

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial included a screening period, up to 5 days active treatment, and follow-up visit. The patients had to visit the trial site up to 3 times.
Pre-assignment Details: 229 patients in total were included
Period: Overall Study
Arm/Group | Angal S (Arm A) | ANTI-ANGIN® FORMULA (Arm B)
Started | 114 | 115
Per Protocol Population | 112 | 111
Safety Population | 114 | 115
ITT Population | 114 | 115
Completed | 114 | 114
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Angal S (Arm A) | ANTI-ANGIN® FORMULA (Arm B) | Total
Number analyzed (Participants) | 114 | 115 | 229
Age, Continuous [Mean (Full Range); unit: Years] | 31.22 [18 to 45] | 30.54 [18 to 50] | 30.88 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 67 | 142
  Male | 39 | 48 | 87
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 114 | 115 | 229

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With a ≥50% TSS Total Score Reduction
Description: Percentage of participants with a ≥50% TSS Total Score Reduction according to the TSS questionnaire completed by the Investigator as compared to the baseline.
  The Tonsillopharyngitis Severity Score (TSS) scale consists of the following symptoms:
  throat pain, difficulty in swallowing, salivation, erythema and fever rated on a 4-point scale (0 = no symptom to 3 = significant symptom). Total score range from 0 - 15.
Time Frame: 4 days
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Angal S (Arm A) | ANTI-ANGIN® FORMULA (Arm B)
Number analyzed (Participants) | 114 | 115
percentage of participants | 96.49 [91.26 to 99.04] | 98.26 [93.86 to 99.79]
Statistical Analysis 1: Comparison: Angal S (Arm A) vs ANTI-ANGIN® FORMULA (Arm B); Test type: Superiority; p = 0.446, Fisher Exact

2. Secondary Outcome: Change From Baseline in TSS Total Score
Description: Change from baseline in TSS total score completed by the Investigator as compared to the baseline.
  The Tonsillopharyngitis Severity Score (TSS) scale consists of the following symptoms:
  throat pain, difficulty in swallowing, salivation, erythema and fever rated on a 4-point scale (0 = no symptom to 3 = significant symptom). Total score range from 0 - 15.
Time Frame: 4 days
Population: ITT population
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Angal S (Arm A) | ANTI-ANGIN® FORMULA (Arm B)
Number analyzed (Participants) | 114 | 115
units on a scale | -6 [-11 to 0] | -6 [-10 to 0]

3. Secondary Outcome: Number of Participants Who Fully Recovered
Description: Number of Participants who Fully Recovered by Day 4 in Group A and by Day 5 in Group B (the outcome of a disease according to the objective evaluation by the Investigator, the total score according to the TSS questionnaire ≤ 2)
Time Frame: Group A: 4 days Group B: 5 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Angal S (Arm A) | ANTI-ANGIN® FORMULA (Arm B)
Number analyzed (Participants) | 114 | 115
Participants | 106 | 107
Statistical Analysis 1: Comparison: Angal S (Arm A) vs ANTI-ANGIN® FORMULA (Arm B); Test type: Superiority; p = 1.0, Fisher Exact

4. Secondary Outcome: Change in the Sore Throat Intensity by 100 mm VAS
Description: Change in the sore throat intensity by 100 mm VAS (visual analogue scale filled in by the patient) at the start and after 3 days of therapy. The VAS is a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." The VAS ranges from 0 to 100. A decrease from baseline in the VAS score to reflect pain intensity indicates a decrease in pain intensity.
Time Frame: 4 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Angal S (Arm A) | ANTI-ANGIN® FORMULA (Arm B)
Number analyzed (Participants) | 114 | 115
mm
  Baseline (Visit 1) | 64.76 (16.29) | 65.84 (18.36)
  Day 4 (Visit 2) | 2.99 (10.33) | 5.06 (11.06)
Statistical Analysis 1: Comparison: Angal S (Arm A) vs ANTI-ANGIN® FORMULA (Arm B); Test type: Superiority; p = 0.145, t-test, 2 sided

5. Secondary Outcome: Period of Time Required for Disappearance of the Disease Symptoms
Description: A period of time required for disappearance of the disease symptoms, determined according to the patient's diary (subjective patient's evaluation), but no more than 5 days during the trial-for patients who have achieved the corresponding outcome.
Time Frame: 5 Days
Population: ITT Population (only cases with disappearance of symptoms within 5 days)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Angal S (Arm A) | ANTI-ANGIN® FORMULA (Arm B)
Number analyzed (Participants) | 114 | 115
Days | 3.75 (0.59) | 3.94 (0.69)
Statistical Analysis 1: Comparison: Angal S (Arm A) vs ANTI-ANGIN® FORMULA (Arm B); Test type: Superiority; p = 0.188, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Percentage of Patients Without Sore Throat According to the Tonsillopharyngitis Severity Score (TSS)
Description: The Tonsillopharyngitis Severity Score (TSS) scale consists of the following symptoms:
  throat pain, difficulty in swallowing, salivation, erythema and fever rated on a 4-point scale (0 = no symptom to 3 = significant symptom). Total score range from 0 - 15.
Time Frame: 4 Days
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Angal S (Arm A) | ANTI-ANGIN® FORMULA (Arm B)
Number analyzed (Participants) | 114 | 115
Percentage of Participants
  Score 0 (no sore throat) | 89.47 | 75.65
  Score 1 | 7.02 | 19.13
  Score 2 | 2.63 | 4.35
  Score 3 | 0.88 | 0.87
Statistical Analysis 1: Comparison: Angal S (Arm A) vs ANTI-ANGIN® FORMULA (Arm B); p1=proportion of patients without sore throat at Day 4 in Arm A p2=proportion of patients without sore throat at Day 4 in Arm B Н0: p1 - p2 ≤ -0.145; Test type: Non-Inferiority — non-inferiority margin 14.5% absolute difference between percentages in group A and B; p = 0.00001, Fisher Exact — p- value for superiority: 0.021; Risk Difference (RD) = 0.14, 95% CI 2-sided [0.03 to 0.24]

ADVERSE EVENTS:
Time Frame: From signing informed consent (Day 1) until completion of the trial (Day 7).
Arm/Group | Angal S (Arm A) | ANTI-ANGIN® FORMULA (Arm B)
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/115
Other Adverse Events (participants affected / at risk) | 7/114 | 11/115
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angal S (Arm A) (N=114) | ANTI-ANGIN® FORMULA (Arm B) (N=115)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 1 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However Novartis does not prohibit any inversdtigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT03095508/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT03095508/SAP_001.pdf